CLINICAL TRIAL: NCT05517512
Title: Low Serum Pregnancy Protein 13 Early in Pregnancy Might Predict the Oncoming Gestational Hypertensive Disorders, Especially Early-onset Preeclampsia
Brief Title: Relation Between Protein 13 and Gestational Hypertensive Disorder
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Amr Sharaf Eldein, Assistant professor of gynecology, Benha University
Other Study IDs: Rc5.6.2022
Record Dates: First submitted 2022-08-09; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Gestational Hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Gestational Hypertension
  Interventions: Diagnostic Test: Estimation of Protein 13
- Pre Eclampsia
  Interventions: Diagnostic Test: Estimation of Protein 13
- Control
  Interventions: Diagnostic Test: Estimation of Protein 13

INTERVENTIONS:
Diagnostic Test: Estimation of Protein 13 — Serum biomarkers' levels were measured using enzyme-linked immunosorbent assay (ELISA) kits according to the manufacturer's instructions and were read using a 96 well microplate ELISA reader (Dynatech. MR 7000)
  1. Human placental growth factor (PLGF) was measured with the enzyme-linked immunoassay (ELISA) kit (catalog no. DPG00 SPG00 PDPG00, R&D Systems Inc., Minneapolis, USA) by quantitative sandwich enzyme immunoassay technique (20).
  2. Human soluble fms-like tyrosine kinase-1 (sFlt-1) was measured with the enzyme-linked immunoassay (ELISA) kit (catalog no. MBS601616, MyBioSource, Inc., California, San Diego, USA) by quantitative sandwich enzyme immunoassay technique (21).
  3. Human pregnancy protein 13 was measured with the enzyme-linked immunoassay (ELISA) kit (catalog no. ab100553, Abcam Inc., Cambridge, USA) by quantitative sandwich enzyme immunoassay technique (22).

SUMMARY:
the attendants of the clinic with a one-missed period (T0) underwent determination of baseline blood pressure (BP) measures and gave blood samples for estimation of levels of placental growth factor (PLGF), soluble fms-like tyrosine kinase-1 (sFlt-1) and pregnancy protein 13 (PP13). The same evaluation was repeated on the 6th, 24th, 32nd, and 36th gestational week (GW). Twenty non-pregnant women gave samples as a negative control group.

ELIGIBILITY:
Inclusion Criteria:

* Normotensive women who attended the clinic with a one-missed period (T0)

Exclusion Criteria:

* History of essential hypertension (HTN)
* renal diseases
* hepatic diseases
* cardiac diseases
* metabolic syndrome
* body mass index (BMI) >35 kg/ m2
* congenital heart diseases

Ages: 21 Years to 33 Years | Sex: Female
Age Groups: Adult
Study Population: Non Hypertensive pregnant women
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2021-03-14 (Actual); Study Completion 2022-03-19 (Actual)

PRIMARY OUTCOMES:
Serum biomarkers and GHD | 9 months
  The primary outcome is the ability of early ELISA estimation of biomarkers for prediction of GHD

CONTACTS AND LOCATIONS:
Locations (1):
- Banha University, Banhā, El- Qalyobia, Egypt